# **Document Coversheet**

Study Title: A randomized, parallel-group open-label trial of ENDS users switching from flavors of potentially high-toxicity profile to flavors of potentially low-toxicity profile (CRoFT\_3.2)

| Institution/Site: | Roswell Park Comprehensive Cancer Center |
|----------------------------------|------------------------------------------|
| Document (Approval/Update) Date: | 05/02/2024 |
| NCT Number: | NCT05423340 |
| IRB Number | I 2588022 |

Protocol #:

Participant Name:

I 2588022

V.2

Participant MR#:

# ROSWELL PARK CANCER INSTITUTE

<u>Title</u>: A Randomized, Parallel-group Open-label Trial of ENDS Users Switching from Flavors of Potentially High-toxicity Profile to Flavors of Potentially Low-toxicity Profile (CRoFT\_3.2)

## **Principal Investigator:**

Maciej Goniewicz. PhD, PharmD Roswell Park Comprehensive Cancer Center Elm and Carlton Street Buffalo, New York 14263 716-845-8541

Roswell Park Study Number: I-2588022

Consent Form Given to Patient Taking Part in an Investigational/Clinical Research Study

#### KEY INFORMATION ABOUT THIS RESEARCH STUDY

This is a research study being done by the doctors at the Roswell Park Comprehensive Cancer Center. Research studies include only those people who choose to take part. Your participation is voluntary. Please take your time to make your decision. Discuss it with your family and with people who are important to you.

We are asking you to take part in this study because you are a current e-cigarette user. As of May 2020, <u>Public Health Law Article 13-F Section 1399-MM-1</u> prohibits the sale of flavored vapor products that do not have an FDA marketing order. Therefore, this policy only prohibits the sale of the products in NYS; possession of the products is not banned or illegal. For this study we will ask information about your current flavor and device use including where you purchase your products. All data provided to us by you will not be disclosed to anyone outside of our research team.

<u>Study Purpose</u>: The purpose of this study is to find out if there is a difference in respiratory symptoms between people who vape different flavors. In addition, this study is also designed to find out if there is a change in respiratory symptoms in people who stop vaping and start using oral nicotine products.

<u>Study Duration and Number of Participants</u>: It is expected this study will take about 3 years or will continue until the needed number of participants are enrolled. We expect to enroll 216 participants from Roswell Park over 3 years.

Your participation in this study will include 4 laboratory study sessions that each last about 45-60 minutes along with a follow-up phone call 30 days after your final laboratory study session.

Laboratory session #2 must occur 7 days after session#1 (±2 days of flexibility). Session #3 must occur 30 days after session #2 (±7 days of flexibility). Lastly, session #4 must take place 60 days after session#3 (±14 days of flexibility). Participants that are unable to make study sessions within the time frame described will be taken off study.

Protocol #: I 2588022
 V.2
Participant Name:
MR#:

**Exams, Tests and Procedures:** This study involves exams, tests and procedures, all of which will be done for research-related purposes.

Listed below are key research-related tests and procedures that you will undergo during the study:

- Your vital signs will be taken at the beginning of every laboratory session.
- You will have blood taken at every session (approximately 9 teaspoons total)
- Females of child-bearing age will be asked to provide a urine sample and be tested for pregnancy during the first session, prior to using the study product.
- You will provide saliva samples.
- You will provide breath samples.
- You will provide an oral rinse sample using mouthwash.
- You will provide a urine sample.
- You will provide nasal samples.
- You may be asked to switch to using a different flavor in your vape or to stop vaping and use an oral nicotine product for 90 days depending on what study group you are placed into.

Section 3 of this document provides additional information on exams, tests and procedures involved with this study. Exams, tests and procedures being done for research-related purposes are required for your participation in the study according to the schedule outlined in Section 3.

<u>Study Costs</u>: There is no cost to participate in this study. You may receive the following products as part of this study depending on which group you are placed into. These products will be provided to you at no cost by the study sponsor (Roswell Park):

- Juul
- Hyde
- Tobacco flavor free-based nicotine solution
- Rogue oral nicotine pouches

Section 9 of this document provides additional information on how to find out what costs are related to this research study.

Side Effects and Risks: While you take part in this study, you may be at risk for side effects from use of the study products, such as nausea, headache, nicotine withdrawal, respiratory or mouth irritation. Another important risk to be aware of is that nicotine overdose may occur from Juul, Rogue, Hyde, and tobacco flavor nicotine solution usage. You should discuss these risks with your doctor/study investigator. It is very important that you notify your doctor/study investigator right away about any side effects, problems, or unusual experiences you may have while on this study. This will decrease the chance that the side effects continue or become worse. Sometimes there are other resources that we can provide to you to make you more comfortable. If severe side effects do develop, you and your doctor/study investigator may decide it is in your best interest to stop taking part in the study.

Section 6 of this document provides more detailed information on possible side effects and risks.

Protocol #:

Participant Name:

I 2588022 V.2

Participant Nam MR#:

**Potential Benefits:** The results and information gained from this study will be used in helping to develop and implement standardized quality procedures for flavored liquids. There is no direct benefit for those who decide to participate and enroll in this study. It is hoped that the study will provide information to guide regulation of tobacco and nicotine products.

<u>Other Options</u>: If you do not join this study, there are no alternative options. If you wish to quit vaping, you should discuss these options with your doctor, a certified tobacco treatment specialist, or contact the New York State Smokers' Quitline (1-866-697-8487).

The type of study, the risks, benefits, discomforts, and other important information about this study are discussed below.

#### ADDITIONAL INFORMATION ABOUT THIS RESEARCH STUDY

It is important that you read and understand the following facts that apply to anyone that takes part in our studies:

- a) This study is considered research. It is investigational.
- b) Taking part in the study is voluntary.
- c) You may withdraw from the study at any time without penalty, loss of any benefits or access to care at Roswell Park to which you are otherwise entitled.
- d) If you should decide not to take part in this study, it will not affect your care at Roswell Park now or in the future.
- e) You may not be helped from taking part in this study, but we may get information that will help others.
- f) If we become aware of important new information that may relate to your willingness to participate in this study we will inform you of this new information.
- g) If you decide to stop being in the study, you should talk with your doctor first about this decision so you are informed whether stopping study participation may have any effects on your health.

#### 1. What is the purpose of this study?

The purpose of this study is to determine for the first time if there if there are any changes in the respiratory system (nose, mouth, throat, bronchia, and lungs) between people who vape flavored e-liquids (such as fruit, candy, dessert, etc.) versus people who switch from using flavored e-liquids to tobacco flavored e-liquids. In addition, this study will also determine if there are any respiratory changes in people who quit vaping flavored e-liquids and start using 'tobacco free' oral nicotine pouches.

This study will also be able to see if people are able to switch flavor use for 90 days while on study or quit vaping and use oral nicotine pouches for the 90 days. We will also assess some biological responses, such as markers of stress, inflammation, and oral health from using the nicotine products. For example, some biomarkers will tell us whether there may be some inflammation in your lungs. The data provided will further scientific knowledge concerning ways to improve the safety of vaporized products and to inform product regulation.

Protocol #:


I 2588022 V.2

Participant Name: MR#:

# 2. What are the study groups?

If you are eligible for the study, you will be randomly placed into 1 of 3 groups:

- If you are placed in <u>Group 1</u>, then you will be asked to continue using your usual flavored e-liquid throughout the whole study.
- If you are placed in <u>Group 2</u>, then you will be asked to switch to tobacco flavored e-liquid, and we will provide you with the e-liquid for the whole study duration.
- If you are placed in <u>Group 3</u>, then we will ask that you stop vaping and switch to using 'tobacco free' oral nicotine pouches that will be provided to you.

Another way to find out what will happen to you during this study is to read the chart below. Start reading at the left side and read across to the right, following the lines and arrows.



This study involves random (by chance) placement into one of the 3 groups. You cannot choose the group you will be placed in. Randomization is a process used to place study participants in different groups. A statistician will use a computer to assign the groups. By using randomization, the groups can be compared objectively. You will have an equal chance of being placed in either of the 3 groups.

## Group 1

If you are placed in Group 1, you will be asked to continue using your usual flavor(s) and to not change flavors during 90 days.

#### Group 2

If you are placed in Group 2 then you will be asked to use a new assigned tobacco flavor regularly for 90 days, and not use any alternative or additional flavors during this time. We will provide you with the tobacco flavored e-liquid that most similarly matches what you are currently vaping at the time of the study. For example:

If you use a MOD device, you will be provided free-based tobacco refill solution 4 mg nicotine. The liquid will be purchased from a local vapor shop in Buffalo, NY (Yeti Vape).

Protocol #: I 2588022
 V.2
Participant Name:
MR#:

If you use a POD device, then we will provide you with a Juul device. The Juul is a pod-style vaping device, with each pod pre-filled with 0.7mL of a nicotine solution. Nicotine solutions will be Virginia tobacco flavored and contain 5.0% nicotine (~50 mg/mL), primarily in the form of nicotine salts (Figure 1).

Figure 1 Juul



If you use a disposable device, then we will provide you with a Hyde device. The Hyde device has a pre-filled 1.6ml tank built in. The solution in the tank contains 5.0% nicotine (~50 mg/mL) and is Gold tobacco flavor (Figure 2).

Figure 2 Hyde



#### Group 3

If you are placed in Group 3, then you will be asked to stop vaping for 90 days and instead only use the provided 'tobacco free' nicotine pouches. Oral nicotine pouches are similar to snus, smokeless tobacco, in that they are portioned pouches designed to be placed between the lip and gum. These pouches do not produce any emissions and are 100% tobacco leaf-free.

For those in Group 3 you will be provided 'tobacco free' ROGUE nicotine pouches. The 3 mg pouches in Mango flavor will be used (Figure 3).

Figure 3 ROGUE



Protocol #:

Participant Name:
MR#:

I 2588022 V.2

## 3. If I take part in this study, what tests and procedures will I have done?

Listed below are the procedures that will be done at each study visit:

- 1. **Respiratory Rate and Pulse Oximetry:** A trained technician will place a sensor on your fingertip to measure the oxygen level in your blood. Then the technician will count the number of complete respiratory cycles (one inhale and one exhale) you breathe in 60 seconds.
- 2. **Expired Breath:** We will measure the amount of carbon monoxide (CO) in your breath to confirm whether you currently smoke cigarettes or other products. This will be done using a portable device called Smokerlyzer® in a similar way as police officers used to measure alcohol in a driver's breath. You will blow into the handheld machine and if it reads over the limit, you will be classified as a current smoker and we will need to exclude you from the study.
- 3. <u>Comprehensive set of questionnaires using a touch screen monitor:</u> You will be given a touch screen monitor with many questions to answer. These questions include information about your health status, lifestyle, work, and use of tobacco products. We will ask you about:
  - a. <u>Demographics</u>, <u>Medical History and Drug Use</u>: **(only at the first visit)** The questions will ask about your demographics (your age, gender, socioeconomic status, drug (including marijuana) and medication use (ever and past 30 day), and diet. If you are a woman, you will also be asked about whether you are pregnant.
  - b. <u>Current and Past Use of Tobacco Products:</u> We will ask whether you currently use or have used various tobacco products
  - c. <u>History of Switching from Tobacco to e-cigarettes</u>: **(only at first visit).** Since you may be an ex-smoker who quit tobacco cigarettes and switched to vaping products, we will ask you how many times you attempted to quit smoking, if you ever used cigarettes and vapor products at the same time and when you totally quit cigarettes and switched completely to vaping products.
  - d. <u>Use of Flavored Product:</u> At each visit we will ask you to estimate and list the different flavors you used in the past month and how much e-liquid or e-juice you approximately used each day.
  - e. <u>Flavor Preference:</u> We will ask you many questions about the various flavors you currently vape or vaped in the past. For example, we will ask you about the very first flavor you used, flavors you use now, flavors you used in the past, and the brands of flavors you used.
  - f. <u>Use of a Regular Brand:</u> We will ask you a series of questions about the brand of e-liquid or e-juice you use.
  - g. <u>Personal History of Respiratory Symptoms/Diseases (past 30-days)</u>: We will ask you questions about your breathing and health since the last study visit (at your first visit, we will ask that you recall your breathing patterns and health 30 days before coming in).

Protocol #: I 2588022
 V.2
Participant Name:
MR#:

- h. Quality of Life as Affected by Respiratory Condition (past 30-days): We will ask you a series of questions about your breathing and how it may affect your daily activities and social life.
- i. <u>Secondhand Exposure:</u> We will ask you to remember if during the past week you were around anyone smoking cigarettes whether in your home, a vehicle, a public place or at work.
- j. <u>House Rules about Vaping and Smoking:</u> We will ask you several questions about vaping in your home.
- k. <u>Oral Health:</u> We will ask you several questions about your oral health and hygiene habits.
- 1. <u>COVID-19</u> Questionnaires: Each month, we will ask you questions about your possible exposure to COVID-19 or any symptoms. In addition, we will be asking you about your personal feelings regarding the virus as well as if you received the vaccination and when you received the vaccine. If you report receiving the vaccine or booster within 7 days of your scheduled study session, we will simply ask that you reschedule your visit 7 days after receiving the vaccine.
- m. <u>Marijuana/Cannabis Use:</u> While you are encouraged to not use any tobacco products and or other drugs while on study, we would like to monitor any marijuana/cannabis use while you are on study.
- n. Subjective Gastrointestinal Symptoms: At every visit we will ask you to fill out the GERD Health-Related Quality of Life Questionnaire in order to monitor any gastrointestinal side effects that might be taking place.
- 4. <u>Collection of Exhaled Breath Condensate (EBC):</u> Study staff will hand you a small tube that you will breathe normal into for about 2 minutes. You will hold the tube to your mouth and blow in and out like you would if you were snorkeling under water. The tube will later be transferred to the lab where we will measure markers of inflammation in your breath.
- 5. <u>Blood Collection:</u> At each study visit, a nurse or trained phlebotomist will collect 7 small vials of blood (approximately 9 teaspoons). We will transfer your blood sample to our lab where we will run numerous tests to measure markers of inflammation. We will also conduct a rapid test using your serum to see if you are positive or negative for COVID-19 antibodies.
- 6. **Spirometry:** We will test your lung function using a handheld device that you will blow into. This breath test will measure the amount of air in your lungs and the time it took to empty it out in one breath. These are indicators of how healthy your lugs are.
- 7. **Nasal Epithelium Brushing:** Trained study staff will use a small sterile brush to take a sample from your nose. Later in the lab, we will look at the cells from your nose to check if these cells change over time or get damaged.
- 8. Exhaled Nitric Oxide(FeNO): This is a hand-held machine that you will simply blow into to measure NO amount. Nitric oxide is another indicator of inflammation in your upper respiratory tract.

Protocol #: I 2588022
 V.2
Participant Name:
MR#:

- 9. <u>Strength of Respiratory Muscles</u>: We will test the strength of your lung muscles using a handheld machine that you will blow into. The machine will measure the strength of your breath as you breathe into it.
- 10. <u>Urine Sample Collection:</u> At each visit, you will be asked to provide a urine sample. We will test your urine sample to identify whether you have been exposed to any toxic chemicals.
- 11. <u>Collection of Product Sample:</u> At each study visit, you will be asked to bring the flavored liquid and vaping products you use or do not use during study visits. We want you to keep all bottles, pods, or devices whether used up or not used up in between sessions. This will help us to keep track of the amount of product you use throughout the study. In our lab, we will measure what flavoring chemicals have been added to your liquid.
- 12. <u>Puffing Topography:</u> At the end of each visit, we will hook your vaping product up to a small device and have you puff as you usually do. The small device will measure how many puffs you take, how long each puff is and the amount of air you puffed. You will be allowed to puff as long as you wish.
- 13. <u>Saliva Sampling:</u> We will ask you to provide a saliva sample at each study visit by chewing on the provided Salivette® swab (similar to a cotton swab used by dentists) for 120 seconds to simulate saliva production.
- 14. <u>Oral rinse samples:</u> At each study visit you will be asked to provide an oral rinse using 10mL(2tsp) of Scope® mouthwash. Collection will involve a 30-second oral rinse broken into three 5-second swish and 5-second gargle sessions, which you will then spit into a sterile collection cup for analysis of the oral bacterial, fungal, and viral microbiome.

Collected urine, plasma, exhaled breath condensate (EBC), and nasal epithelium samples will be de-identified and sent to the Biomarkers, Genomics & Epigenomics (BGE) Core located at the University of Rochester Medical Center in Rochester, New York for study analysis purposes only.

#### 4. Will I be informed of research results?

If we learn new information from research tests or analyses during this study that may be important to your health, we will share that information with you. Such information will be provided to you by the study staff.

To maintain the integrity of this research study, you will not have the right to review or copy your study results related to this research until the study is complete. At the conclusion of the research study, and at your request, you may have access to summarized published results of the study.

# 5. Why would I be taken off the study early?

You may be taken off the study for any of the following reasons:

- Your medical condition changes
- New information becomes known to us that would influence your decision to remain on the study
- The sponsor of the study, Roswell Park, may decide to stop or change the study
- You do not follow the study schedule or requirements

Protocol #:

Participant Name:
MR#:

I 2588022 V.2

- You experience unacceptable side effects
- You no longer want to participate

## 6. What risks and discomforts are involved?

While you take part in this study, you may be at risk for side effects. Overall, there is minimal risk for serious adverse reactions as a consequence of enrolling in this study. Any side effects are expected to resolve shortly after the study. The side effects may be mild, moderate, or severe. Many side effects go away shortly after stopping, but occasionally, side effects can be serious, long lasting, or may be permanent.

It is not possible to tell which side effect will affect you or how mild or severe the side effect might be. We can only tell you what other people have experienced.

It is very important that you notify your doctor right away about **any** side effects, problems, or unusual experiences you may have while on this study. You can also call the study nurse with the phone number that will be provided to you at the start of the study. This will decrease the chance that side effects continue or become worse. Sometimes there are other resources that we can provide to make you more comfortable. If severe side effects do develop, you and the study investigator/physician may decide it is in your best interest to stop taking part in the study.

The study products used in this study may cause all, some, or none of the side effects listed.

The risks and side effects for NICOTINE are listed below.

<u>Very likely Side Effects</u>: In 100 people who use nicotine products, approximately more than 50 experienced the following:

- Nicotine withdrawal; including sadness, anxiety, irritability, anger, difficulty concentrating, appetite change, weight gain, insomnia, and decreased heart rate.
  - O You may experience nicotine withdrawal while on study if you are placed in Group 2 or Group 3 because you will be asked to stop using your regular nicotine product and start using a different nicotine product that we will provide you. Therefore, there is a small chance that your body may not get the exact same amount of nicotine you are used to getting while using your regular nicotine product.

<u>Less likely Side Effects:</u> In 100 people who use nicotine products, approximately 10-19 experienced the following:

- Nicotine overdose; including nausea, sleep disturbance, headache, and vomiting.
  - You may experience nicotine overdose while on study if you are placed in Group 2 or Group 3 because you will be asked to stop using your regular nicotine product and start using a different nicotine product that we will provide you. Therefore, depending on how often you use the provided nicotine product, your body may get a larger amount of nicotine than it is used to getting from your regular nicotine product. The likelihood of this happening is very small.
- Respiratory irritation; including irritation of the mucosal membranes of the upper respiratory tract.

Protocol #:  Participant Name: I 2588022 V.2

MR#:

• Mouth irritation; irritation of the mucosal membranes of the mouth (inner lip, gum).

# **Risks from Tests/Procedures:**

- **Blood Draw:** there is a small risk of local pain, swelling, bruising, or infection. Significant complications (beyond typical local pain and mild bruising) are expected to be uncommon.
- **Nasal swabs:** there may be minor nasal irritation.
- Emotional distress: participants may experience psychological discomfort during assessments when discussing feelings and attitudes about vaping and/or using nicotine products.
- Inconvenience: participants may experience inconvenience due to multiple study visits required.
- Respiratory Irritation: Some people who vape may experience irritation of the mucosal membranes of the upper respiratory tract (i.e., the membranes that line your mouth and throat), but since you vape on a regular basis, we do not think that this is likely to occur.

We will exclude you or postpone procedures if you demonstrate chronic or acute respiratory problems.

#### 7. Reproductive risks:

This study may involve risks to you or your unborn child that are not known at this time therefore, you should not become pregnant while you are participating in this study. Also, you should not nurse your baby while on this study. Women of childbearing potential will be required to take a pregnancy test before being allowed to take part in this study. The pregnancy test must be negative before you enter this study.

Women of childbearing potential will be asked to practice an effective method of birth control while on this study and for a time after the second session. Please discuss this with your doctor.

When you sign this consent form, to the best of your knowledge, you are not pregnant and do not plan to become pregnant while taking part in this study. Should you become pregnant during this study, you need to immediately tell your study doctor and obstetrician. If you wish you may request a referral for counseling or ask about counseling (such as genetic counselor, social worker, or psychologist.) to discuss this further.

#### 8. What are my responsibilities in this study?

If you choose to take part in this study you will need to:

- Keep your study appointments. While on study you are expected to:
  - o Come in for Session#2 7 days after session#1 (+/-2 days of flexibility) In other words you can come to Session#2 no earlier than 5 days since Session#1 and no later than 9 days after Session#1. It is very important to adhere to these specified times for each study session.
  - O Session #3 must occur 30 days after session #2 (+/-7 days of flexibility).

Protocol #: I 2588022
 V.2
Participant Name:
MR#:

- Lastly, session #4 must take place 60 days after session#3 (+/-14 days of flexibility).
- Do not smoke cigarettes or use other tobacco products or drugs, such as marijuana, throughout the study duration.
- Tell study staff about:
  - o All medications and supplements you are taking
  - Any side effects
  - O Any changes in your product use (i.e. if you start using a new vaping product and/or liquid, or if you do not adhere to the study product given to you while on study)
  - o If you stop vaping and/or using the study products.
- Keep the study products out of the reach of children and do not share the study products with any other person.

# 9. What happens if I am injured as a result of this study?

If you believe you have been injured as a direct result of your participation in this research study, notify the Roswell Park Patient Advocate at (716) 845-1365 or the Study Doctor at (716) 845-5412.

Medical diagnosis and treatment for the injury will be offered, and a determination will be made regarding appropriate billing for the diagnosis and treatment of the injury. A financial counselor can be reached at 716-845-3161 to provide an explanation of coverage and to answer questions you may have regarding study related billing.

You do not give up any legal rights by signing this form. You are not prevented from seeking to collect compensation for injury related to malpractice, fault, or blame on the part of those involved in the research.

#### 10. Will I be paid for joining this study?

You will receive the following payment for participating in this study:

<u>All participants</u> will be paid <u>\$400</u> for completing all 4 visits. An additional \$20 will be given for the completion of the follow-up phone call 1 month after Session#4 is complete. Cash will be given after each session is complete as follows:

Table 1. Cash compensation given to all participants

| ARM | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Follow-Up |
|----------|---------|-------------|---------|---------|-----------|
| 1, 2 & 3 | \$50 | <b>\$75</b> | \$125 | \$150 | \$20 |

It is possible that this research project may result in developing devices, new drugs, or procedures that could be used for commercial profit by the sponsor or other entities. If this happens, you understand that you will not receive any financial payment or share in any commercial profit for

Protocol #:  Participant Name: MR#:

I 2588022 V.2

the use of your information and biospecimens (such as blood or tissue samples) collected as part of this research.

# 11. Where can I find more information?

If you wish to stop vaping and or stop the use of any nicotine products, you can call the New York State Smokers Quitline at 1-866-697-8487 (1-866-NY-QUITS) or visit www.nysmokefree.com.

## 12. Who do I contact with questions?

You are free to ask questions at any time about this study and to ask for more information from the doctor identified on this document. If you have any questions, concerns or complaints about this study, you should contact the study doctor identified on the first page of this document. In case of an emergency after regular hospital hours, you should telephone (716) 845-2300 and ask for the doctor on call. You are also able to reach out to the study nurse at any point while on study. A number will be provided to you at your first study session.

If you have questions about your rights as a research subject or you feel you have been injured as a result of your participation in this research study, you can call the Roswell Park Patient Advocate (Support) Office at (716) 845-1365. You should also feel free to contact the Patient Advocate Office at any time while considering participation, during participation or once your participation is complete. This office is unaffiliated with any specific research study. They can help you obtain additional information regarding your research participation and your rights as a research subject or how to proceed should you feel you have been injured as a result of your participation. They are available to discuss any problems, concerns, questions or input you may have.

It may be necessary to contact you at a future date regarding new information about this research study. For this reason, we ask that you notify the Patient Access office at 716-845-1049 or stop at the Registration Desk in the Lobby of Roswell Park to update us of any change in your address.

#### What about confidentiality?

Your privacy is very important to us and the researchers will make every effort to protect it. Your information collected in this study may be given out if required by law. For example, certain states require doctors to report to health boards if they find a disease like tuberculosis. However, the researchers will do their best to make sure that any information that is released will not identify you. Some of your information, and/or information about your specimen, from this study will be kept in a central database for research. Your name or contact information will not be put in the database.

There are organizations that may inspect the study records and your information. These organizations are required to make sure your information is kept private, unless required by law to provide information. Some of these organizations are:

- The study sponsor, Roswell Park Cancer Institute
- The Institutional Review Board, IRB, is a group of people who review the research with the goal of protecting the people who take part in the study.
- The Food and Drug Administration and the National Cancer Institute in the U.S., and similar ones if other countries are involved in the study.

Protocol #:  Participant Name: I 2588022 V.2

MR#:

Information that does or can identify you may be removed from your information or biospecimens (such as blood or tissue samples) so that it may be used or disclosed for other purposes, including use for future research studies or distributed to another investigator for future research studies without additional informed consent from you or your legally authorized representative.

# **Certificate of Confidentiality**

As an additional measure to protect your privacy, a Certificate of Confidentiality has been issued from the United States Government, National Institutes of Health, for this study. With this Certificate, the investigators and institutions involved in this study cannot be forced to disclose information that may identify you, even by a court subpoena, in any federal, state, or local civil, criminal, administrative, legislative, or other proceeding. We will use this Certificate to resist any demands for information that would identify you, with the following exceptions:

- The Certificate cannot be used to resist a request for your information from the United States Government when the information is to be used for auditing or evaluation of federally funded projects or for information that must be disclosed to meet the requirements of the Food and Drug Administration (FDA).
- State law requires we report cases of diseases that spread easily, or abusive behavior (toward a child, a partner, or an elderly person), and people who say they are going to hurt themselves or someone else.
- The Certificate does not prevent you or a member of your family from voluntarily releasing information about yourself or involvement in this research. Also, if you have given written consent to an insurer, employer, or other person to receive research information, then we may not use the Certificate to withhold the information.

#### **Genetic Information Protection**

A Federal law, called the Genetic Information Nondiscrimination Act (GINA), generally makes it illegal for health insurance companies, group health plans, and most employers to discriminate against you based on your genetic information. This law generally will protect you in the following

- Health insurance companies and group health plans may not request your genetic information that we get from this research.
- Health insurance companies and group health plans may not use your genetic information when making decisions regarding your eligibility or premiums.
- Employers with 15 or more employees may not use your genetic information that we get from this research when making a decision to hire, promote, or fire you or when setting the terms of your employment.

GINA's prohibitions apply to 'genetic information' which is defined as including receipt of genetic services (genetic tests, genetic counseling, or genetic education) by an individual or family member participating in clinical research.

GINA does not protect you against genetic discrimination by companies that sell life, disability or long-term care insurance.

Roswell Park and the researchers involved in this study will not reveal the results of your genetic tests to health insurers or employers and your records will be kept confidential to the extent described in this consent form.

Protocol #:  Participant Name: I 2588022 V.2

MR#:

#### **OPTIONAL RESEARCH**

This part of the consent form is about optional studies that you can choose to take part in. You will not get health benefits from any of these studies. The research from these studies may help other people with cancer or other diseases in the future. You can still take part in the main study even if you say "no" to this optional research.

We would like to store leftover samples of blood, saliva, nasal epithelium, exhaled breath condensate, and oral samples that we get during the tests/procedures done as part of the study. If you agree, these samples may be kept in a specimen bank here at Roswell Park.

The samples will be labeled so your name and your identity will remain unknown to the researchers. It is not possible for us to know now all the different ways the samples may be studied in the future. We would also like to store information collected on you in this clinical study including your age, and ethnic background.

Information from studies using your samples and your medical information will be collected along with information from other people who volunteer for this optional research. Researchers can request to study the samples and medical information stored in the specimen and data bank.

This includes researchers at Roswell Park as well as from other universities, the government, and drug or health-related companies in the United States or other countries. Information from studies of your samples and your medical information might also be shared broadly by placing the information into one or more large scientific databases maintained at Roswell Park or at other institutions or by the federal government where it is stored along with information from many other people and from other studies. Researchers can request to study the combined information to learn more about cancer or other diseases. Some information from these large databases may be made freely available to the public (unrestricted access) but will not contain any information specific to you or any other participant. Information from studies using your samples and your medical information may also be put in a controlled-access database in which researchers need to get permission to use the information for a research project. Researchers who are approved to access the information in the controlled-access database will need to agree not to attempt to identify you.

We will not give researchers information that could directly identify you. We will take many steps to protect the privacy of people who take part. We will remove your name and any other information that could directly identify you from your samples and information. We will replace the direct identifiers with a code number and only certain study staff will have access to the key that will link the code number to your identity. By protecting your identity in this manner, researchers who study your samples and information will not know who you are. There is a risk that someone could get access to the data we have stored about you. It is also possible that the information from your genome, when combined with information from other public sources could be used to identify you. We believe the chance of this happening is very small but we cannot make guarantees. Your privacy and the confidentiality of your information are very important to us and we will make every effort to protect them.

It is not possible for us to know now what tests will be discovered in the future. We cannot give you a list of all the possible ways the sample will be used. We are asking that you give your permission for us to take, store and do research on the sample without contacting you again in the

Protocol #:

Participant Name:

I 2588022 V.2

Participant No MR#:

future. It is possible that future research projects may result in developing treatments, devices, new drugs, or procedures that could be used for commercial profit. If this happens, you understand that you will not receive any financial payment or share in any commercial profit for the use of your biospecimens (such as blood or tissue samples) that had been stored for future research.

If you give permission for the sample now and change your mind later, you will need to write to the doctor listed on the first page of this form and let him/her know that you changed your mind. If we have not already used the sample, it will be destroyed and not used. If you have any questions, please ask your doctor.

Consenting to have your remaining samples stored is not needed to take part in the rest of the study. If you decide not to join in this part of the study, you can still join the rest of the study. Any amounts remaining from the samples provided after running all specified study analyses will be destroyed and tested no further.

I agree that someone from Roswell Park Comprehensive Cancer Center may contact me in the future to ask me to take part in more research.

| PLEASE CHECK ONE BOX | |
|---|---|
| YES | NO |
| My leftover blood can be used in research. PLEASE CHECK ONE BOX | |
| YES | NO |
| My leftover saliva, breath, and nasal cell samples can be used in research. PLEASE CHECK ONE BOX | |
| VES | NO |

Protocol #:  Participant Name: I 2588022

V.2

CRS registration Medical Records

MR#:

# **Statement of Investigator/Person Conducting the Informed Consent Discussion:**

I certify that the nature and purpose, the potential benefits and possible risks associated with participation in this research study have been explained and that any questions about this information have been answered. A signed copy of this consent will be given to the participant.

| SIGNATURE | DATE | TIME |
|---|---|---|
| PRINTED NAME | | |
| Participant's Statement of Consent: | | |
| By signing below, you agree that: | | |
| <ul> <li>You have been told of the reasons for this stud</li> </ul> | y. | |
| • You have had the study explained to you. | 1 . 1 1. | |
| • You have had all of your questions answer | ed, including | those about areas you did not |
| <ul><li>understand, to your satisfaction.</li><li>You have carefully read this consent form and</li></ul> | will receive a | signed copy of this form |
| <ul> <li>You do <b>not</b> waive any <b>legal</b> rights you have un</li> </ul> | | |
| <ul> <li>You willingly give your consent to voluntarily</li> </ul> | | |
| Participant: | | |
| SIGNATURE | _DATE | TIME |
| PRINTED NAME | | |
| Witness Signature is needed in the following cir Not Applicable The person consenting cannot write – mark mu The person consenting cannot read - consent has The person consenting cannot understand interpreted. (The witness should be fluent in both English as | st be made as<br>as been read to<br>English and | appropriate. o him/her. the consent has been verbally |
| Witness Statement: | | |
| The person consenting has signed this document in | my presence | ·. |
| SIGNATUREDAT | E | TIME |
| PRINTED NAME | | CONSENT HANDLING Original to CRA-Regulatory with Race Ethnicity if applicable |
| RELATIONSHIP TO PARTICIPANT | | Copy to: Patient |
| | | Fatient |